CLINICAL TRIAL: NCT02631928
Title: Single-center, Randomized, Double-blind, 2-treatment, 2-period Crossover Trial in Healthy Subjects to Demonstrate PK Bioequivalence and to Compare the PD Properties of Julphar Insulin 30/70 and Huminsulin® Profil III
Brief Title: Pharmacokinetic (PK) Bioequivalence and Pharmacodynamics (PD) of Julphar Insulin 30/70 and Huminsulin® Profil III
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Julphar Gulf Pharmaceutical Industries (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: INSULCT002; 2015-003993-34 (EudraCT Number)
Record Dates: First submitted 2015-11-25; First posted 2015-12-16 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: biphasic human insulin; biosimilar
MeSH Terms: conditions — Diabetes Mellitus | interventions — biphasic human insulin 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Julphar Insulin 30/70 (Experimental): human biphasic insulin, 100 IU/mL, single subcutaneous injection of 0.6 IU/ kg body weight
  Interventions: Drug: human biphasic insulin
- Huminsulin® Profil III (Active Comparator): human biphasic insulin, reference, 100 IU/mL, single subcutaneous injection of 0.6 IU/ kg body weight
  Interventions: Drug: human biphasic insulin, reference

INTERVENTIONS:
Drug: human biphasic insulin — investigational insulin, biosimilar human insulin suspension of 30% normal insulin and 70% basal protamined insulin
  Other Names: Julphar Insulin 30/70
  Arms: Julphar Insulin 30/70
Drug: human biphasic insulin, reference — marketed product, human insulin suspension of 30% normal insulin and 70% basal (NPH) insulin
  Other Names: Huminsulin® Profil III
  Arms: Huminsulin® Profil III

SUMMARY:
This study in healthy volunteers aims to demonstrate similar PK and PD properties of the new human biphasic insulin, Julphar Insulin 30/70 and an already approved reference insulin, Huminsulin® Profil III. All participants will receive both study treatments on two separate dosing days.

DETAILED DESCRIPTION:
Daily injections of insulin is a necessity for many patients with diabetes mellitus in order to treat hyperglycaemia. Julphar Insulin 30/70 and Humininsulin® Profil III are both biphasic insulins, i.e. consist of a mixture of short-acting soluble insulin and intermediate-acting isophane insulin. The new insulin, Julphar Insulin 30/70, is biosimilar to Huminsulin® Profil III. Demonstration of similar absorption (PK) and effects (PD) are necessary to achieve market approval of Julphar Insulin 30/70.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedures that would not have been performed during normal management of the subject).
* Healthy male subject.
* Age between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 28.0 kg/m^2, both inclusive.
* Fasting plasma glucose concentration <= 100 mg/dL.

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs or related products.
* Previous participation in this trial. Participation is defined as randomised.
* Receipt of any medicinal product in clinical development within 3 months before screening.
* Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator.
* Any history or presence of clinically relevant cardiovascular, pulmonary, respiratory, gastrointestinal, hepatic, renal, metabolic, endocrinological haematological, dermatological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness as judged by the Investigator.
* Surgery within 12 weeks before the start of the study or blood donation of more than 500 mL (or considerable blood loss) or plasma donation within the last 3 months.
* Increased risk of thrombosis, e.g., subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
* Clinically significant abnormal values for haematology, biochemistry, coagulation, or urinalysis as judged by the Investigator.
* Supine blood pressure (BP) at screening (after resting for 5 minutes in a supine position) outside the range of 90 to 140 mmHg for systolic BP or 50 to 90 mmHg for diastolic BP (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial) and/or resting supine pulse < 50 beats per minute.
* Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
* Any disease or condition that, in the opinion of the Investigator, would represent an unacceptable risk for the subject's safety.
* Positive to the screening test for Hepatitis Bs antigen or Hepatitis C antibodies and/or a positive result to the test for HIV-1/2 antibodies or HIV-1 antigen.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (prescription and non-prescription drugs) within 14 days before first trial drug administration and/or anticoagulant therapy, with the exception of stable treatment with thyroid hormones, paracetamol and ibuprofen for occasional use to treat pain.
* Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 21 units of alcohol per week (one unit of alcohol equals about 330 mL of beer, one glass of wine of 120 mL, or 40 mL spirits).
* A positive result in the alcohol and/or urine drug screen at the screening visit.
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) who is not able or willing to refrain from smoking and use of nicotine substitute products 1 day before and during the inpatient period.
* Subject with mental incapacity or language barriers precluding adequate understanding or cooperation or who, in the opinion of the Investigator, should not participate in the trial.
* Potentially noncompliant or uncooperative during the trial, as judged by the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
PK: AUCins.0-24, harea under the serum insulin concentration curve from 0-24 hours | 24 hours
PK: Cins.max, maximum observed insulin concentration | 24 hours
  24 hours

SECONDARY OUTCOMES:
PK: AUCins.0-6h, AUCins.0-12, areas under the serum insulin concentration curve in the indicated time intervals | 12 hours
PK: AUCins.0-∞, area under the serum insulin concentration-time curve from 0 hours to infinity | 24 hours
PK: tmax, time to maximum observed serum insulin concentration | 24 hours
PK: t½, terminal serum elimination half-life calculated as t½=ln2/λz | 24 hours
PK: λz, terminal elimination rate constant of insulin | 24 hours
PD: AUCGIR.0h-last, area under the glucose infusion rate curve from 0 hours until the end of clamp | 24 hours
PD: GIRmax, maximum observed glucose infusion rate | 24 hours
PD: AUCGIR.0-6h, AUCGIR.0-12h, areas under the glucose infusion rate curve in the indicated time-intervals | 12 hours
PD: tGIR.max, time to maximum glucose infusion rate | 24 hours
PD: Onset of action, time from trial product administration until blood glucose concentration has decreased at least 5 mg/dL from baseline | 24 hours
  baseline is defined as the mean of blood glucose levels from -6, -4, and -2 minutes before trial product administration as measured by the glucose clamp device
Adverse events | from the first trial drug administration until the final examination
  Through study completion, approx.up to approx. 39 days for each subject and up to 6 month for total study duration..
Local tolerability findings | dosing period, approx.up to 39 days for each subject
  at the injection site. Through study completion,
  The local tolerability at the injection site will be evaluated by means of the following assessments:
  * spontaneous pain
  * pain on palpation
  * itching
  * erythema
  * oedema
  * induration/infiltration
  * other Each of these assessments will be reported on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe). The evaluation and the actual time of the assessment will be recorded.
Laboratory safety parameters | from screening until final examination, approx.up to 60 days for each subject
  Including haematology, biochemistry and coagulation including serology (only at screening) parameters. Through study completion,
Physical examination findings | from screening until final examination, approx.up to 60 days for each subject
  Through study completion,
Changes in vital signs | from screening until final examination, approx.up to 39 days for each subject
  Through study completion,
Changes in Electrocardiogram recordings | from screening until final examination, approx.up to 60 days for each subject
  Through study completion,

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany